CLINICAL TRIAL: NCT05868304
Title: Dynamic and Isometric Strength Analyses of Lower Extremity Blood Flow Restriction Training: A Randomized Controlled Trial
Brief Title: Lower Extremity BFR-randomized Controlled Trial Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Orr Limpisvasti, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002454
Record Dates: First submitted 2023-03-01; First posted 2023-05-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Blood Flow Restriction (BFR); Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Standard strengthening group (no BFR) (Active Comparator): Participants will warm up on a stationary bike for 5 minutes
  The program will consist of the following exercises using a 30,15,15,15 rep scheme:
  Banded squats Step ups (8 inch) Romanian dead lifts (RDL)
  Interventions: Other: Stanard strengthening program.
- Group 2 - Low-load BFR group (Experimental): Participants will warm up on a stationary bike for 5 minutes BFR will be applied to non-dominant limb (dominant limb is determined as the preferred leg for kicking a ball)
  The program will consist of the following exercises using a 30,15,15,15 rep scheme:
  Banded squats Step ups (8 inch) Romanian dead lifts (RDL)
  Interventions: Device: BFR; Other: Stanard strengthening program.

INTERVENTIONS:
Device: BFR — Exercises may involve warm up on a stationary bike for 5 minutes, application of a BFR cuff (a cuff that often uses air to inflate around a limb) on the selected extremity, and exercise sets (e.g. banded squats, step ups, Romanian dead lifts). We will record metrics on an iPad. Testing will be done with ForceDecks and ForceFrames (system for measuring muscle strength and imbalance).
  Arms: Group 2 - Low-load BFR group
Other: Stanard strengthening program. — The exercise program will be completed 3 times per week Participants will warm up on a stationary bike for 5 minutes
  The program will consist of the following exercises using a 30,15,15,15 rep scheme:
  Banded squats Step ups (8 inch) Romanian dead lifts (RDL)

SUMMARY:
The purpose of this research is to determine the effects of low-load blood flow restriction (BFR) training compared to conventional strengthening using dynamic force plate and isometric force frame analyses in healthy subjects.

DETAILED DESCRIPTION:
The purpose of this research is to determine the effects of low-load blood flow restriction (BFR) training compared to conventional strengthening using dynamic force plate and isometric force frame analyses in healthy subjects. The primary research procedures are:

Subjects will be randomized into either BFR or conventional strengthening groups.

BFR and conventional strengthening programs will be implemented. Force plate and force frame data will be collected at baseline, 4, 6, 8, 12, and 16 weeks.

Subject Population. The study will enroll 18 healthy volunteers. The study includes 6 visits.

The total study duration for each subject is 16 weeks.

The device the investigators intend to use is Class I and in a class of devices that is exempt from the FDA requirement for premarket notification/approval (exempt from 510K or PMA), which would not be "subject to section 510(k), 515, or 520(m) of the Federal Food, Drug, and Cosmetic Act

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers without history of knee pathology requiring physical therapy or surgery
* Individuals between 18 and 40 years old

Exclusion Criteria:

* History of venous thromboembolism or other hematologic disorder Pregnant
* Coronary artery disease, peripheral arterial disease, or hypertension (> 140/90 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
The change in Force plate measures from baseline to 16 weeks | Measured at 4, 6, 8, 12, and 16 weeks.
  Force (N)
The change in Force plate measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Power (W)
The change in Force plate measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Velocity M/Se
the changes in Force plate measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Relative strength index (RSI)
the change in Force plate measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Displacement
the changes in Force Frame measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Force (N)
the changes in Force Frame measures from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  power (W)
the changes in Force Frame measure from baseline to 16 weeks | Measured at 4,6,8,12 and 16 weeks.
  Velocity M/sec

CONTACTS AND LOCATIONS:
Locations (1):
- Cedar Sinai Kerlan jobe orthopedic institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No